CLINICAL TRIAL: NCT04139811
Title: Evaluation of Primary Internal Limiting Membrane Peeling in Cases of Rhegmatogenous Retinal Detachment
Brief Title: Evaluation of Visual Functions After Pars Plana Vitrectomy With and Without Internal Limiting Membrane Peeling in RRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hossam Mohamed Moharram, Assistant professor of ophthalmology, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 66-7/2018
Record Dates: First submitted 2019-09-24; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Retinal Detachment
Keywords: Internal limiting membrane; multifocal electoretinogram (ERG); OCT-Angiography
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-ILM peeling group (Other): vitrectomy without ILM peeling is done to all cases
  Interventions: Other: Pars Plana Vitrectomy
- ILM peeling group (Other): vitrectomy with ILM peeling is done to all cases
  Interventions: Other: Pars Plana Vitrectomy

INTERVENTIONS:
Other: Pars Plana Vitrectomy — vitrectomy with and without ILM peeling

SUMMARY:
Internal limiting membrane peeling is performed during vitrectomy for macular diseases such as macular holes, macular edema due to diabetic retinopathy and retinal vein occlusion.

The incidence of epiretinal membrane formation after vitrectomy for rhegmatogenous detachment has been reported to range from 4.4% to 12.8%.

In this study, the efficacy and safety of internal limiting membrane peeling will be studied in vitrectomy for rhegmatogenous retinal detachment and if it is essential to peel it in those cases or not.

DETAILED DESCRIPTION:
interventional observational study comparing vitrectomy with versus without internal limiting membrane peeling in cases of rhegmatogenous retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* All eyes with recent macula-off rhegmatogenous retinal detachment (RRD).

Exclusion Criteria:

* Complicated cases with advanced proliferative vitreoretinopathy (PVR).
* Patients with retinal vascular disorders and other macular disorders.
* Combined tractional and rhegmatogenous detachment.
* Previous retinal reattachment surgery or Intravitreal injections.
* Glaucomatous patients.
* Patients with corneal opacity which impairs good visualization.

Ages: 20 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
anatomical outcome | 6 months follow up
  Rate of retinal reattachment using indirect ophthalmoscopy
epiretinal membrane | 6 months follow up
  incidence rate of epiretinal membrane formation after surgery in % percent

SECONDARY OUTCOMES:
functional outcome | 6 months follow up
  visual functions using log Mar Best Corrected Visual Acuity (BCVA)
superficial capillary density | 6 months follow up
  measurement of percent (%) of superficial and deep capillary density using Optical Coherance Tomography Angiography
multi-focal Electroretinogram | 6 months follow up
  measurement of P1 amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Othman, MD, Principal Investigator — sub-investigator; Ahmed Shawkat, MD, Principal Investigator — sub-investigator; khalid Murad, Principal Investigator — sub-investigator; Mohamed Abdullah, Principal Investigator — sub-investigator
Locations (1):
- Minia UNiversity hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdullah ME, Moharram HEM, Abdelhalim AS, Mourad KM, Abdelkader MF. Evaluation of primary internal limiting membrane peeling in cases with rhegmatogenous retinal detachment. Int J Retina Vitreous. 2020 May 7;6:8. doi: 10.1186/s40942-020-00213-4. eCollection 2020. PMID 32411388